CLINICAL TRIAL: NCT02195037
Title: Changes in Cardiac Output During Delayed Umbilical Cord Clamping
Status: Completed | Type: Observational
Sponsor: Sharp HealthCare (Other)
Responsible Party: Principal Investigator, Anup Katheria, M.D., Director of Neonatal Research, Sharp HealthCare
Other Study IDs: CO-DCC
Record Dates: First submitted 2014-07-17; First posted 2014-07-21 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2014-08

CONDITIONS: Cardiac Output, Low
Keywords: Delayed Cord Clamping
MeSH Terms: conditions — Cardiac Output, Low

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Recently, the American College of Obstetricians and Gynecologists (ACOG) recommended a delay of 30-60 seconds in umbilical cord clamping for all newborn infants. This delay allows the newborn to receive his/her own blood from the placenta (placental transfusion) which helps their transition in the first hours of life. The purpose of the study is to learn about the amount of blood flow to and from the baby's heart during normal newborn transition

ELIGIBILITY:
Inclusion Criteria:

* Healthy full term infants
* Delivered by vaginal birth
* Estimated gestational age of 37+0to 41+6 weeks corrected gestational age

Exclusion Criteria:

* Multiples
* Known fetal anomalies (including cardiac defects).
* Instrumentation during delivery (forceps or vacuum)
* Non-reducible nuchal cord during delivery.
* Any maternal or neonatal indication requiring immediate cord clamping.

Max Age: 1 Minute | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Healthy full term infants delivered by vaginal birth with an estimated gestational age of 37+1 to 41+6 weeks corrected gestational age
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-07; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Cardiac Output | 5 minutes of Life

SECONDARY OUTCOMES:
Stroke Volume | 5 Minutes of Life
Bilirubin level | until discharge
Hemoglobin level | until discharge

CONTACTS AND LOCATIONS:
Overall Officials: Anup Katheria, MD, Principal Investigator — Sharp HealthCare
Locations (1):
- Sharp Mary Birch Hospital for Women and Newborns, San Diego, California, United States

REFERENCES:
- [Derived] Katheria AC, Wozniak M, Harari D, Arnell K, Petruzzelli D, Finer NN. Measuring cardiac changes using electrical impedance during delayed cord clamping: a feasibility trial. Matern Health Neonatol Perinatol. 2015 May 22;1:15. doi: 10.1186/s40748-015-0016-3. eCollection 2015. PMID 27057332